CLINICAL TRIAL: NCT00572871
Title: Hormonal and Bone Turnover Marker Response to an Acute Bout of Resistance or Plyometric Exercise
Status: Completed | Type: Observational
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Sponsor
Other Study IDs: 1097239; 65438 (Other: University of Missouri)
Record Dates: First submitted 2007-12-12; First posted 2007-12-13 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-09

CONDITIONS: Osteoporosis; Osteopenia
MeSH Terms: conditions — Osteoporosis; Bone Diseases, Metabolic | interventions — Plyometric Exercise; Resistance Training

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — serum plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Exercise after fasting: Will complete 2 resistance exercise sessions and 2 plyometric exercise sessions after a 10-hour fast
  Interventions: Other: resistance exercise
- No exercise: Will complete a ten-hour fast but do no exercise
  Interventions: Other: No exercise
- Exercise after snack: Will complete 2 resistance exercise sessions and 2 plyometric exercise sessions 2 hours following a 500 calorie nutritional supplement
  Interventions: Other: plyometric exercise

INTERVENTIONS:
Other: plyometric exercise — single bout of plyometric exercise
  Groups: Exercise after snack
Other: resistance exercise — single bout of resistance exercise
  Groups: Exercise after fasting
Other: No exercise — Will not do any exercise
  Groups: No exercise

SUMMARY:
We are interested in determining if there exist a short-term response in the serum markers and hormones that participate in the regulation of bone tissue formation and breakdown to a single, high-intensity exercise session of weight lifting (resistance exercise) or jumping (plyometrics). We are also interested in determining if the bone marker response to exercise is altered by changing the negative energy state caused by the exercise treatment, when subjects are given a moderate calorie meal.

DETAILED DESCRIPTION:
Bone tissue responds to impact and strain forces, like high-intensity exercise, by upregulating the bone remolding process, resulting in the deposition of calcium phosphate minerals into the collagen matrix of bone. Bone remodeling is a continually active process that involves both activation cells regulating bone formation (osteoblasts) and resorption (osteoclasts). Alterations in the balance between formation and resorption are critical for changes in bone density and mineral content to occur, which is regulated by several hormones including vitamin D and growth hormone, the sex hormones estrogen and testosterone, and parathyroid hormone. Importantly, it remains unclear how single bouts of physical activity contribute to the overall changes in remodeling and whether those acute alterations can be detected in the hours after exercise. Additionally, research studies examining the effects of exercise on bone remodeling often draw blood samples after 24 hours of physical inactivity, potentially diminishing the magnitude of the exercise response. Therefore, we plan to evaluate the acute effects of plyometrics and resistance exercise on changes in serum hormones and markers of bone turnover in non-sedentary, healthy males, with or without a moderate calorie supplement.

ELIGIBILITY:
Inclusion Criteria:

* Male
* No symptoms of disease
* Non-sedentary
* Age 25-65

Exclusion Criteria:

* Medications or supplements that affect bone metabolism or prevent exercise
* Previous or current medical condition affecting bone health, including osteoporosis.
* Cardiovascular disease
* Metallic implants affecting accuracy of bone density scan
* Current smoker
* Current participation in high-intensity jumping or resistance exercise in the last 3 months.

Ages: 25 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Male participants apparently healthy and non-sedentary free of disease that affects bone and not have used or currently use any medication that affects bone.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2007-12; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
serum bone turnover markers | 24 hours

SECONDARY OUTCOMES:
serum hormones regulating bone turnover | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Pamela S Hinton, Ph.D., Principal Investigator — University of Missouri-Columbia

IPD SHARING:
Plan to Share IPD: No